CLINICAL TRIAL: NCT03723200
Title: Treatment of Obstetric Hemorrhage With Fibrinogen and Blood Products: Retrospective Analyzes
Brief Title: Analyzes of Hemorrhagic Obstetric Patients Whose Were Used Fibrinogen
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ayca Sultan Sahin, Principal Investigator, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2018.9.19
Record Dates: First submitted 2018-10-24; First posted 2018-10-29 (Actual); Last update posted 2018-10-30 (Actual); Status verified 2018-10

CONDITIONS: Hemorrhage
Keywords: Hemorrhagic; Obstetric; Fibrinogen
MeSH Terms: conditions — Hemorrhage | interventions — Fibrinogen

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

INTERVENTIONS:
Other: Fibrinogen and blood products — Fibrinogen and blood products

SUMMARY:
The files of hemorrhagic obstetric patients undergoing surgery and followed in the intensive care unit and using Fibrinogen and blood products were included in the study between January 2015- September 2018 at the Anesthesiology and Reanimation Clinic of SBU Kanuni Sultan Süleyman Training and Research Hospital. Patients under 18 years of age were excluded from the study. In this study, ages, operation types, number of blood and products, the amount of fibrinogen, the results of the hemogram and bleeding parameters, the levels of fibrinogen, the duration of hospital stay and the intensive care unit were recorded.

DETAILED DESCRIPTION:
Bleeding is an important event that threatens the patient's life. Too much blood and blood products can be used in massive bleeding. However, unwanted allergic reactions may occur in blood and blood product transfusions. Fibrinogen is the first coagulation factor in coagulopathy. Some studies have shown that when the fibrinogen level falls to <150-200 mg / dl, the bleeding increases dramatically.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients, underwent surgery and followed in ICU
* Used Fibrinogen and Blood products
* Over 18 years age

Exclusion Criteria:

* Under 18 years age
* Obstetric patients, underwent surgery but not used Fibrinogen and Blood products

Ages: 18 Years to 50 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — obstetric patients
Study Population: - Obstetric patients who underwent surgery and followed in ICU and Used Fibrinogen and Blood products in peroperatively or postoperatively
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Measurement of fibrinogen (mg/L) | 24 hours
  Significant independent predictor for evolution to severe PPH was plasma fibrinogen level.
Measurement of hemoglobin (g/dL) | 24 hours
  Postpartum hemorrhage (PPH) is a major contributor to maternal death and severe maternal morbidity
Amount of fibrinogen consantrates | 24 hours
  in order to avoid PPH
Amount of blood products (unit) | 24 hours
  degree of hemorrhagie

SECONDARY OUTCOMES:
Hospital stay days | 24 hours
  for the recovery time of patients

CONTACTS AND LOCATIONS:
Overall Officials: Ayca Sultan Sahin, MD, Principal Investigator — Kanuni Sultan Suleyman Education and Training Hospital
Locations (1):
- Kanuni Sultan Suleyman Education and Training Hospital, Istanbul, Kucukcekmece, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided